CLINICAL TRIAL: NCT07293390
Title: Mass Balance Study of TQ05105
Brief Title: A Clinical Trial of Mass Balance of [14C] TQ05105 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-I-05
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mass Balance of [14C] TQ05105 in Healthy Chinese Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ05105 (Experimental): Take the [14C]TQ05105 suspension under fasting conditions, ensuring the entire dose is administered within 5 minutes. The total water volume used for drug preparation and administration is approximately 240 mL.
  Interventions: Drug: TQ05105

INTERVENTIONS:
Drug: TQ05105 — Janus Kinase 2 (JAK2) inhibitor

SUMMARY:
To analyze radioactivity excretion and pharmacokinetics in healthy subjects after a single oral dose of [¹⁴C]TQ05105, identifying excretion routes, major metabolites, and biotransformation pathways. Secondary: To determine pharmacokinetics of TQ05105 and metabolites (e.g., TQ12550) via Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS) and assess treatment safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male;
* Age: 18-45 years (inclusive);
* Body weight: Body mass index (BMI) between 19-26 kg/m² (inclusive), with a minimum body weight of 50 kg;
* Voluntarily signs the informed consent form;
* The subject is able to communicate well with the investigator and able to complete the trial in accordance with the protocol requirements.

Exclusion Criteria:

* Abnormalities with clinical significance detected in comprehensive physical examination, routine laboratory tests (complete blood count, blood biochemistry, coagulation function, urinalysis, fecal routine), thyroid function, 12-lead electrocardiogram, chest CT, abdominal ultrasound (liver, gallbladder, pancreas, spleen, kidneys), etc.;
* Abnormal vital signs that remain abnormal upon retesting;
* Abnormalities with clinical significance in ophthalmic examinations (slit-lamp, intraocular pressure, and fundus photography);
* Positive results for Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibody IgG (Anti-HCV IgG), human immunodeficiency virus antibody (HIV-Ag/Ab), or syphilis antibody;
* Positive nucleic acid test result for Coronavirus Disease 2019 (COVID-19);
* Use of any drugs known to inhibit or induce hepatic drug-metabolizing enzymes within 30 days prior to screening (see Appendix 1 for details);
* Use of any prescription drugs, over-the-counter medications, Chinese herbal health products, or dietary supplements (e.g., vitamins, calcium supplements) within 14 days prior to screening;
* History or presence of clinically significant diseases affecting the musculoskeletal, neuropsychiatric, endocrine, circulatory, respiratory, digestive, urinary, or reproductive systems, as judged by the investigator;
* Any medical condition that increases the risk of elevated blood glucose, such as a history of primary diabetes, steroid-induced diabetes, other secondary diabetes, acute or chronic pancreatitis, deemed clinically significant by the investigator;
* History of organic heart disease, heart failure, myocardial infarction, angina, unexplained arrhythmia, torsades de pointes, ventricular tachycardia, atrioventricular block, or long QT syndrome (or related symptoms/family history), deemed clinically significant by the investigator;
* History of interstitial lung disease, severely impaired lung function, severe pulmonary fibrosis, radiation pneumonitis, drug-induced lung disease, or evidence of active pulmonary inflammation on screening chest CT, deemed clinically significant by the investigator;
* Major surgery within 6 months prior to screening or incomplete wound healing; major surgery includes procedures with significant bleeding risk, prolonged general anesthesia, open biopsy, major traumatic injury, or surgery affecting drug absorption, distribution, metabolism, or excretion; or planned surgery during the study;
* History of drug, environmental, or food allergies, allergic constitution, or potential allergy to the investigational drug or its excipients, as judged by the investigator;
* Hemorrhoids or perianal diseases with regular/active bleeding, irritable bowel syndrome, or inflammatory bowel disease;
* Factors affecting oral administration or drug absorption (e.g., swallowing difficulties, gastrointestinal resection, ulcerative colitis, symptomatic/inflammatory bowel disease, intestinal obstruction, etc.);
* Habitual constipation or diarrhea;
* Lactose intolerance (history of diarrhea after consuming milk);
* Alcohol abuse or regular alcohol consumption within 6 months prior to screening (>14 units per week; 1 unit = 360 mL beer, 45 mL 40% spirits, or 150 mL wine); inability to abstain during the trial, or positive alcohol breath test (>0 mg/100 mL) at screening;
* Smoking >5 cigarettes daily within 3 months prior to screening or habitual use of nicotine products, and inability to abstain during the trial;
* Drug abuse or use of soft drugs (e.g., marijuana) within 3 months prior to screening, or hard drugs (e.g., cocaine, amphetamines, phencyclidine) within 1 year prior to screening; or positive urine drug screen at screening;
* Habitual consumption of grapefruit juice or excessive tea, coffee, and/or caffeine-containing beverages, and inability to abstain during the trial;
* Occupation involving long-term exposure to radiation conditions; or significant radiation exposure within 1 year prior to the trial (≥2 chest/abdominal CT scans or ≥3 other X-ray examinations); or prior participation in radioactive drug-labeled trials;
* History of needle or blood phobia, difficulty with blood collection, or inability to tolerate venipuncture;
* Participation in other clinical trials involving investigational drugs or devices within 3 months prior to or during screening, or planned participation during this study; or non-personal participation in clinical trials;
* Vaccination within 1 month prior to screening or planned vaccination during the trial;
* Plans for reproduction or sperm donation during the trial or within 1 year after completion, or unwillingness to use strict contraception during and within 1 year after the trial (see Appendix 3 for details);
* Blood loss or donation ≥400 mL within 3 months prior to screening, or blood transfusion within 1 month prior to screening;
* Other reasons deemed by the investigator to make the subject unsuitable for participation, or voluntary withdrawal by the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
loss rate | From 24 hours prior to administration to 504 hours post-administration
  Total radioactive recovery rate and cumulative total radioactive recovery rate in excreta (urine and feces) for each time interval.
Peak concentration (Cmax) | Before administration, 0.16, 0.33, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after administration
  Maximum plasma drug concentration
Area under drug time curve (AUC0-∞) | Before administration, 0.16, 0.33, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after administration
  Area under the plasma concentration-time curve from time 0 extrapolated to infinite time

SECONDARY OUTCOMES:
Adverse event rate | From before the first administration to 7 days after the administration
  Incidence and severity of adverse events and serious adverse events, and abnormal laboratory examination indicators.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangnan University Affiliated Hospital, Wuxi, Jiangsu, China